CLINICAL TRIAL: NCT05205109
Title: A Phase I/Ib, Multi-center, Open-label, and Dose-finding Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of ATG-037 Monotherapy and Combination Therapy With Pembrolizumab in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of ATG 037 Monotherapy and Combination Therapy With Pembrolizumab in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Antengene Therapeutics Limited (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Antengene Corporation (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATG-037-001; KEYNOTE-E73 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2025-06-09 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATG-037+Keytruda(Pembrolizumab, MK-3475) (Experimental): Part I: Dose Escalation Phase of ATG-037 Monotherapy PartII: Dose Escalation Phase and Dose Expansion Phase of ATG-037 in Upfront Combination with Keytruda(Pembrolizumab, MK-3475)
  Interventions: Drug: ATG-037; Drug: KEYTRUDA ®( Pembrolizumab)

INTERVENTIONS:
Drug: ATG-037 — Part I : ATG-037 will be administered orally once a day (QD) on D-2, then multiple doses of ATG-037 will be administered orally BID for every day from C1D1. A treatment cycle will be defined as 21 days.
  Part II: ATG-037 will be administered orally BID for every day from C1D1.
Drug: KEYTRUDA ®( Pembrolizumab) — Part I: After 2 cycles of ATG-037 monotherapy, eligible participants will receive ATG-037 combination therapy with Keytruda ®(Pembrolizumab) 200mg/Q3W fixed dose for up to 35 administrations (approximately 2 years).
  Part II: Keytruda ®(Pembrolizumab) will be administered from C1.
  Other Names: MK-3475

SUMMARY:
This is a study of ATG-037 Monotherapy and Combination Therapy with Pembrolizumab in Patients with Locally Advanced or Metastatic Solid Tumors

DETAILED DESCRIPTION:
This is a Phase I, Multi-center, Open-label, and Dose-finding Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of ATG-037 Monotherapy and Combination Therapy with Pembrolizumab in Patients with Locally Advanced or Metastatic Solid Tumors.

Number of subjects :

1. 39-51 subjects for Dose escalation phase part 1
2. Maximum of 18 subjects or Dose escalation phase part 2
3. 24-34 subjects per Dose expansion cohort

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study-specific procedures, sampling, and analyses.
2. Aged at least 18 years as of the date of consent.
3. Unresectable Stage III or Stage IV melanoma patients, who have had disease progression on or after at least one prior ICI containing treatment. Patients with mucosal and uveal melanoma types are to be excluded.
4. There is at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
5. Estimated life expectancy of a minimum of 12 weeks.
6. Subjects with acquired immune checkpoint inhibitors resistance (objective response or SD>6 months).
7. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 at ICF signature.
8. Females should be using adequate contraceptive measures until 180 days after the end of treatment, should not be breastfeeding.
9. Male subjects should be willing to use barrier contraception, ie condoms, for the duration of the study and 180 days after the final dose of study treatment.
10. Subjects should have adequate organ function.

Exclusion Criteria:

1. Primary central nervous system disease, central nervous system metastatic disease, leptomeningeal disease, metastatic cord compression or carcinomatous meningitis.
2. Prior exposure to a CD73 inhibitor/antibody or adenosine receptor inhibitor.
3. Patients considered to have rapidly progressive disease (from the starting of prior line therapy to disease progression lasting no more than 90 days).
4. Prior therapy with any chemotherapy, immunotherapy, anticancer agents or investigational products from a previous clinical study within 28 days of the first dose of study treatment or within a period during which the investigational product or systemic anticancer treatment has not been cleared from the body.
5. Radiotherapy with a wide field of radiation within 28 days, or radiotherapy with a limited field of radiation for palliation within 14 days of the first dose of study treatment. Subject must have recovered from all radiation related toxicity, not requiring corticosteroids.
6. Prior major surgery (excluding placement of vascular access) within 28 days of the first dose of study treatment or minor surgical procedures ≤7 days.
7. Except for alopecia, platinum-induced peripheral neurotoxicity (≤Grade 2). Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE 5.0) Grade 1 at the time of ICF signature.
8. Received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher irAE (except endocrine disorders that can be treated with replacement therapy) or was discontinued from that treatment due to Grade 2 myocarditis or recurrent Grade 2 pneumonitis.
9. Subjects receiving unstable or increasing doses of corticosteroids.
10. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension defined as a blood pressure (BP) ≥160/100 mmHg despite medical therapy, unstable or uncompensated respiratory and renal disease, active bleeding diseases, allogeneic stem cell transplantation, or any solid organ transplant, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and server adverse events | One year after last patient first dose
  Will be graded according to the NCI-CTCAE Grading Scale version 5.0.
DLT | Up to 21 Days
  Number of Participants with Dose Limiting Toxicity
MTD | Up to 21 Days
  Maximum tolerated dose of ATG-037
RP2D | Up to 21 Days
  Recommended phase 2 dose of ATG-037

SECONDARY OUTCOMES:
Plasma concentration of ATG-037 and derived PK parameters | One year after last patient first dose
  To characterize the PK/PDx of ATG-037
Inhibition of CD73 enzymatic activity in plasma | One year after last patient first dose
  To evaluate the preliminary antitumor activity of ATG-037 monotherapy and combination therapy with pembrolizumab
ORR as per RECIST v1.1 and DOR, DCR, PFS, OS evaluated by the investigators | One year after last patient first dose
  To evaluate the preliminary antitumor activity of ATG-037 monotherapy and combination therapy with pembrolizumab

OTHER OUTCOMES:
Expression of related biomarkers in archived tumor tissue by IHC | One year after last patient first dose
  To explore potential PDx markers and characterize changes of the immune microenvironment following treatment with ATG-037
Changes in soluble CD73 concentration in serum | One year after last patient first dose
  To explore potential PDx markers and characterize changes of the immune microenvironment following treatment with ATG-037
The number and activation status of immune cells in peripheral blood | One year after last patient first dose
  To explore potential PDx markers and characterize changes of the immune

CONTACTS AND LOCATIONS:
Overall Officials: Ganessan Kichenadasse, MD, Principal Investigator — Southern Oncology Clinical Research Unit; Yi-Long Wu, PhD, Principal Investigator — Guangdong Provincial People's Hospital; Qing Zhou, Principal Investigator — Guangdong Provincial People's Hospital
Locations (7):
- Australia (5):
  - Calvary Mater Newcastle, Sydney, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - One Clinical Research Pty Ltd, Mount Pleasant, Western Australia
- China (2):
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong